

#### CLINICAL STUDY PROTOCOL

**Study Title:** A Phase 3 Randomized Study to Evaluate the Safety and Antiviral

Activity of Remdesivir (GS-5734<sup>TM</sup>) in Participants with Severe

COVID-19

**Sponsor:** Gilead Sciences, Inc.

333 Lakeside Drive Foster City, CA 94404

**IND Number:** 147753

**EudraCT Number:** 2020-000841-15

Clinical Trials.gov

**Identifier:** NCT04292899

**Indication:** COVID-19

**Protocol ID:** GS-US-540-5773

**Contact Information:** The medical monitor name and contact information will be provided

on the Key Study Team Contact List.

**Protocol Version/Date:** Original: 24 February 2020

Amendment 1.0: 15 March 2020 Amendment 2.0: 20 March 2020 Amendment 3.0: 12 April 2020

This study will be conducted under US Food & Drug Administration IND regulations (21 CFR Part 312); however, sites located in the European Economic Area and Switzerland are not included under the IND and are considered non-IND sites.

### **CONFIDENTIALITY STATEMENT**

The information contained in this document, particularly unpublished data, is the property or under control of Gilead Sciences, Inc., and is provided to you in confidence as an investigator, potential investigator, or consultant, for review by you, your staff, and an applicable Institutional Review Board or Independent Ethics Committee. The information is only to be used by you in connection with authorized clinical studies of the investigational drug described in the protocol. You will not disclose any of the information to others without written authorization from Gilead Sciences, Inc., except to the extent necessary to obtain informed consent from those persons to whom the drug may be administered.

# TABLE OF CONTENTS

| TAE | BLE O | F CONTENTS | 2 |
|---|---|---|---|
| LIST | Γ OF I | N-TEXT TABLES | 4 |
| PRO | тосо | OL SYNOPSIS | 5 |
| GLC | OSSAF | RY OF ABBREVIATIONS AND DEFINITION OF TERMS | 10 |
| 1. | INTR | RODUCTION | 13 |
| 1. | | | |
| | 1.1.<br>1.2. | Background | |
| | 1.2. | 1.2.1. General Information | |
| | | 1.2.2. Preclinical Pharmacology and Toxicology | |
| | 1.3. | Rationale for This Study | |
| | 1.4. | Rationale for Dose Selection of Remdesivir | |
| | | 1.4.1. Pediatric Dosing | |
| | 1.5. | Risk/Benefit Assessment for the Study | |
| | 1.6. | Compliance | |
| 2. | ODII | ECTIVES | 10 |
| 2. | | | |
| 3. | STUI | DY DESIGN | 20 |
| | 3.1. | Endpoints | 20 |
| | 3.2. | Study Design | |
| | 3.3. | Study Treatments | |
| | 3.4. | Duration of Treatment. | |
| | 3.5. | Discontinuation Criteria | |
| | 3.6. | End of Study | |
| | 3.7. | Post Study Care | |
| 4. | SUB. | JECT POPULATION | 23 |
| | 4.1. | Number of Subjects and Subject Selection | 22 |
| | 4.1. | 4.1.1. Subject Replacement | |
| | 4.2. | Inclusion Criteria. | |
| | 4.3. | Exclusion Criteria. | |
| 5. | INVE | ESTIGATIONAL MEDICINAL PRODUCTS | 25 |
| | 5.1. | Randomization, Blinding, and Treatment Codes Access | 25 |
| | | 5.1.1. Randomization | |
| | | 5.1.2. Blinding | |
| | 5.2. | Description and Handling of Remdesivir | |
| | | 5.2.1. Formulation | |
| | | 5.2.2. Packaging and Labeling | |
| | | 5.2.3. Storage and Handling | |
| | 5.3. | Dosage and Administration of Remdesivir | |
| | 5.4. | Accountability for Investigational Medicinal Product | 26 |
| | | 5.4.1. Investigational Medicinal Product Return or Disposal | |
| | 5.5. Prior and Concomitant Medications | | |
| 6. | STUI | DY PROCEDURES | 28 |
| | 6.1. | Subject Enrollment and Treatment Assignment | 28 |
| | 6.2. | Pretreatment Assessments. | |
| | 0.2. | 6.2.1. Screening Visit | |

| | | 6.2.2. Baseline/Day 1 Assessments | 29 |
|---|---|---|---|
| | 6.3. | Daily Study Assessments (Days 2-14) | 30 |
| | 6.4. | Additional Assessments | 30 |
| | 6.5. | Day 28 Follow up Assessment (±5 Days) | 30 |
| | 6.6. | Clinical Laboratory Assessments | 31 |
| | <u>6.7.</u> | Physical Examination. | 32 |
| | CCI | | |
| | 6.9. | Ordinal Scale | 32 |
| | 6.10. | Post-treatment Assessments | |
| | 6.11. | Assessments for Early Discontinuation from Study | |
| | | 6.11.1. Criteria for Discontinuation of Study Treatment | |
| | 6.12. | End of Study | |
| | 6.13. | Post Study Care | |
| | 6.14. | Sample Disposition and Storage (Non-PK Samples) | 34 |
| | CCI | | |
| 7. | ADVI | ERSE EVENTS AND TOXICITY MANAGEMENT | 35 |
| | 7.1. | Definitions of Adverse Events and Serious Adverse Events | 25 |
| | /.1. | 7.1.1. Adverse Events | |
| | | 7.1.2. Serious Adverse Events | |
| | 7.2. | Assessment of Adverse Events and Serious Adverse Events | |
| | 7.2. | 7.2.1. Assessment of Causality for Study Drugs and Procedures | |
| | | 7.2.2. Assessment of Severity | |
| | 7.3. | Investigator Requirements and Instructions for Reporting Adverse Events and Serious | |
| | , | Adverse Events. | 37 |
| | | 7.3.1. Requirements for Collection Prior to Study Drug Initiation | |
| | | 7.3.2. Adverse Events | |
| | | 7.3.3. Serious Adverse Events | 37 |
| | 7.4. | Gilead Reporting Requirements | 38 |
| | 7.5. | Clinical Laboratory Abnormalities and Other Abnormal Assessments as Adverse Events or | |
| | | Serious Adverse Events | |
| | 7.6. | Special Situations Reports | |
| | | 7.6.1. Definitions of Special Situations | |
| | | 7.6.2. Instructions for Reporting Special Situations | 40 |
| 8. | STAT | ISTICAL CONSIDERATIONS | 42 |
| | 8.1. | Analysis Objectives and Endpoints | |
| | | 8.1.1. Analysis Objectives | |
| | | 8.1.2. Primary Endpoint | |
| | | 8.1.3. Secondary Endpoint | |
| | 8.2. | Planned Analyses | |
| | 0.2. | 8.2.1. Interim Analysis | |
| | | 8.2.2. Primary Analysis | |
| | | 8.2.3. Final Analysis | |
| | 8.3. | Analysis Conventions. | |
| | 0.01 | 8.3.1. Analysis Sets | |
| | | 8.3.2. Data Handling Conventions | |
| | 8.4. | Demographic and Baseline Characteristics Analysis | |
| | 8.5. | Efficacy Analysis | |
| | | 8.5.1. Primary Analysis | |
| | | 8.5.2. Secondary Analyses | 45 |
| | 8.6. | Safety Analysis | 45 |
| | | 8.6.1 Extent of Exposure | 45 |

| | | 8.6.2. | Adverse Events | 45 |
|---|---|---|---|---|
| | | 8.6.3. | Laboratory Evaluations | 46 |
| | CCI | | | |
| | 8.8. | • | nents for Multiplicity | |
| | 8.9. | | Size | |
| | 8.10. | Data M | onitoring Committee | 47 |
| 9. | RESP | ONSIBIL | ITIES | 48 |
| | 9.1. | Investig | gator Responsibilities | 48 |
| | | 9.1.1. | Good Clinical Practice | 48 |
| | | 9.1.2. | Financial Disclosure | 48 |
| | | 9.1.3. | Institutional Review Board/Independent Ethics Committee Review and Approval | 40 |
| | | 9.1.4. | Informed Consent (or Assent) | |
| | | 9.1.4. | Confidentiality | |
| | | 9.1.5. | Study Files and Retention of Records | |
| | | 9.1.0. | · | |
| | | 9.1.7. | Case Report Forms | |
| | | | Investigator Inspections. | |
| | 9.2. | 9.1.9. | Protocol Compliance | |
| | 9.2. | 9.2.1. | * | |
| | | 9.2.1. | Protocol Modifications | |
| | 0.2 | | Study Report and Publications | |
| | 9.3. | 9.3.1. | vestigator/Sponsor Responsibilities | |
| | | | Payment Reporting | |
| | | 9.3.2. | Access to Information for Monitoring | |
| | | 9.3.3. | Access to Information for Auditing or Inspections | |
| | | 9.3.4. | Study Discontinuation | |
| 10. | REFE | RENCES | | 53 |
| 11. | APPE | NDICES | | 54 |
| | | ndix 1. | Investigator Signature Page | |
| | | ndix 2. | Study Procedures Table | |
| | Apper | ndix 3. | Pregnancy Precautions, Definition for Female of Childbearing Potential, and | |
| | | | Contraceptive Requirements | 57 |
| | | | LIST OF IN-TEXT TABLES | |
| | Table | 1. | Data Entry Requirements When Only One Result of Multiple Results Is Recorded | |
| | | | for a Given Day | 32 |

#### PROTOCOL SYNOPSIS

Gilead Sciences, Inc. 333 Lakeside Drive Foster City, CA 94404

| <b>Study Title:</b> | A Phase 3 Randomized Study to Evaluate the Safety and |
|---------------------|-------------------------------------------------------|
|---------------------|-------------------------------------------------------|

Antiviral Activity of Remdesivir (GS-5734<sup>TM</sup>) in Participants

with Severe COVID-19

**IND Number:** 

**EudraCT Number:** 

**Clinical Trials.gov Identifier:** 

147753

2020-000841-15

NCT04292899

### **Study Centers Planned:**

Up to approximately 160 centers globally

### **Objectives:**

The purpose of this study is to provide remdesivir (RDV) to participants with severe COVID-19.

The primary objective of this study is as follows:

 To evaluate the efficacy of 2 RDV regimens with respect to clinical status assessed by a 7-point ordinal scale on Day 14

The secondary objective of this study is as follows:

To evaluate the safety and tolerability of RDV

### **Study Design:**

This is a Phase 3 randomized, open-labeled, multi-center study of RDV therapy in participants with severe COVID-19.

The study will be conducted in two parts. In Part A, approximately 400 participants who meet all eligibility criteria and who are not mechanically ventilated may be randomized in a 1:1 ratio into one of the following treatment groups:

**Treatment Group 1:** continued standard of care therapy together with IV RDV 200 mg on Day 1 followed by IV RDV 100 mg on Days 2, 3, 4, and 5

**Treatment Group 2:** continued standard of care therapy together with IV RDV 200 mg on Day 1 followed by IV RDV 100 mg on Days 2, 3, 4, 5, 6, 7, 8, 9, and 10

Part B will enroll participants on mechanical ventilation and, after enrollment to Part A is complete, any additional participants. In Part B, up to an additional approximately 5600 participants who meet all of the eligibility criteria will be enrolled, based on whether they are mechanically ventilated at enrollment, to receive:

**Mechanically Ventilated Treatment Group:** continued standard of care therapy together with IV RDV 200 mg on Day 1 followed by IV RDV 100 mg on Days 2, 3, 4, 5, 6, 7, 8, 9, and 10

**Extension Treatment Group:** continued standard of care therapy together with IV RDV 200 mg on Day 1 followed by IV RDV 100 mg on Days 2, 3, 4, 5, 6, 7, 8, 9, and 10

If the 5-day dosing regimen used in Treatment Group 1 of Part A is selected for Part B, all participants in the Extension Treatment Group and all new participants will be reassigned to receive treatment for a total of 5 days. National and local regulatory authorities will be informed.

Participants in Part A of the study will be the primary efficacy population. Participants enrolled in Part B will have data reported descriptively at study completion.

Number of Subjects Planned:

Approximately 6000

Target Population:

Participants with severe COVID-19

**Duration of Treatment:** 

The duration of treatment with RDV will be up to 10 days

Diagnosis and Main Eligibility Criteria: Participants with COVID-19 confirmed by polymerase chain reaction (PCR) who meet the following criteria:

- Willing and able to provide written informed consent, or with a legal representative who can provide informed consent, or enrolled under ICH E6(R2) 4.8.15 emergency use provisions as deemed necessary by the investigator (age ≥18), or willing and able to provide assent (age ≥12 to <18, where locally and nationally approved) prior to performing study procedures</li>
- Hospitalized
- SpO<sub>2</sub>  $\leq$  94 % on room air or requiring supplemental oxygen at screening
- Radiographic evidence of pulmonary infiltrates

Study Procedures/ Frequency: At screening, after the participant has provided informed consent or assent, demographic and baseline characteristics, medical history, and concomitant medications will be documented. Vital signs including temperature, respiratory rate, and SpO<sub>2</sub> will be recorded. Radiographic imaging will be performed if not already available. SARS-CoV-2 testing by PCR testing will be performed; if this testing has been performed within the previous 4 days, no repeat testing is required.

If safety laboratory results from the screening day are not already available, laboratory testing including alanine aminotransferase (ALT) and aspartate aminotransferase (AST), serum creatinine, and creatinine clearance will be performed according to local practice.

In Part A, after screening procedures, eligible participants will be randomized into 1 of the 2 treatment groups in a 1:1 ratio to receive:

**Treatment Group 1:** continued standard of care therapy together with IV RDV 200 mg on Day 1 followed by IV RDV 100 mg on Days 2, 3, 4, and 5

**Treatment Group 2:** continued standard of care therapy together with IV RDV 200 mg on Day 1 followed by IV RDV 100 mg on Days 2, 3, 4, 5, 6, 7, 8, 9, and 10

In Part B, after screening procedures, eligible participants will be assigned to receive:

**Mechanically Ventilated Treatment Group:** continued standard of care therapy together with IV RDV 200 mg on Day 1 followed by IV RDV 100 mg on Days 2, 3, 4, 5, 6, 7, 8, 9, and 10

**Extension Treatment Group:** continued standard of care therapy together with IV RDV 200 mg on Day 1 followed by IV RDV 100 mg on Days 2, 3, 4, 5, 6, 7, 8, 9, and 10 as determined by review of the data. Treatment may be reduced to a total of 5 days following analysis of the data from Part A.

The date of randomization will be considered Day 1 and all participants randomized to receive RDV should receive their initial dose on Day 1.

On study Days 1 through 14 or until discharge, whichever is earlier, 7-point ordinal scale of clinical status, vital signs including respiratory status will be measured and adverse events (AEs) and concomitant medications will be documented. Laboratory testing will be performed according to SOC practice with results for white blood cell count, hemoglobin and/or hematocrit, platelets, creatinine, creatinine clearance, glucose, total bilirubin, ALT, AST, and any SARS-CoV-2 testing being reported to the Sponsor.

In addition, even if not performed as standard of care, white blood cell count, hemoglobin and/or hematocrit, platelets, creatinine, creatinine clearance, glucose, total bilirubin, ALT, AST will be performed at Days 1, 3, 5, 8, 10, and 14 or until discharge, whichever is earlier.



Test Product, Dose, and Mode of Administration:

Remdesivir (GS-5734) for injection, 100 mg, for IV administration

Reference Therapy, Dose, and Mode of Administration:

None

Criteria for Evaluation:

Safety: Incidence of treatment-emergent AEs and treatment-emergent

clinical laboratory abnormalities

Efficacy: Clinical status assessed by a 7-point ordinal scale on Day 14

#### **Statistical Methods:**

The primary endpoint will be analyzed using a proportional odds model. The null hypothesis being tested is whether the odds of improvement on the ordinal scale is the same for the two treatment groups (i.e., whether the common odds ratio is equal to 1). The odds ratio and 95% confidence interval will be provided.

Treatment-emergent AEs and laboratory abnormalities will be summarized using descriptive statistics and listed by subject.



### Sample Size:

In Part A, a total of approximately 400 participants will be randomized in a 1:1 ratio to 2 groups (200 participants per group)

A sample size of 400 participants (200 participants in each group) achieves > 85 % power to detect an odds ratio of 1.75 using a two-sided significance level of 0.05.

The sample size for Part B is based on the anticipated need for RDV and current trends in the COVID-19 epidemic.

This study will be conducted in accordance with the guidelines of Good Clinical Practice (GCP) including archiving of essential documents.

### GLOSSARY OF ABBREVIATIONS AND DEFINITION OF TERMS

°F Fahrenheit
AE adverse event

ALT alanine aminotransferase AST aspartate aminotransferase

AUC<sub>tau</sub> area under plasma concentration-time curve over dosing interval

BLQ below the limit of quantitation

CDC Centers for Disease Control and Prevention

CoV Coronavirus
CRF case report form

CRO contract/clinical research organization

CSR clinical study report

d deciliter

DAIDS Division of AIDS

DMC data monitoring committee

EBOV Ebola virus

eCCGs eCRF Completion Guidelines eCRF electronic case report form EDC electronic data capture

EGFR epidermal growth factor receptor eSAE Electronic Serious Adverse Event

EU European Union

EudraCT European Clinical Trials Database

FAS Full Analysis Set

FDA Food and Drug Administration FSH follicle-stimulating hormone

g grams

GCP Good Clinical Practice

Gilead Gilead Sciences

HIV human immunodeficiency virus

HLGT high-level group term HLT high-level term

IB investigator's brochure

ICH International Conference on Harmonisation (of Technical Requirements for Pharmaceuticals

for Human Use)

IDMC independent data monitoring committee

IEC independent ethics committee
IND investigational new drug
IRB institutional review board

IUD intrauterine device

IV intravenous

IWRS interactive web response system

J Joule kg kilogram

LAM lactational amenorrhea method LLOQ lower limit of quantitation

LLT lower-level term

LPV lopinavir

LPV/RTV-IFNb LPV/RTV + interferon-beta

MARV Marburg virus

MedDRA Medical Dictionary for Regulatory Activities

MERS Middle East Respiratory Syndrome

min minute

NHPs nonhuman primates
OAT organic anion transporter

PBMC peripheral blood mononuclear cell
PBPK physiologically-based pharmacokinetic

PCR polymerase chain reaction

PK pharmacokinetic(s)
PT preferred term

PVE Pharmacovigilance and Epidemiology

QT electrocardiographic interval between the beginning of the Q wave and termination of the T

wave, representing the time for both ventricular depolarization and repolarization to occur

RDV remdesivir

RNA ribonucleic acid

RSV respiratory syncytial virus RT reverse transcriptase

RTV ritonavir

SADR serious adverse drug reaction

SAE serious adverse event

SARS Severe Acute Respiratory Syndrome
SBECD sulfobutylether β-cyclodextrin sodium

SDV source data verification SOC system organ class

SOP standard operating procedure

SUSAR suspected unexpected serious adverse reaction

TM test method

ULN upper limit of normal

US United States

V-A ECMO Veno-arterial extracorporeal membrane oxygenation

V-V ECMO Veno-venous extracorporeal membrane oxygenation

WHO World Health Organization

### 1. INTRODUCTION

# 1.1. Background

In December 2019, a series of pneumonia cases of unknown cause emerged in Wuhan, Hubei, China. Sequencing analysis from the patients' respiratory tract samples indicated a novel coronavirus (CoV), which was named COVID-19. As of 23 February 2020, more than 78,000 confirmed cases have been identified in Wuhan, other provinces in China, and in multiple countries outside China {World Health Organisation (WHO) 2020}. More than 2400 deaths associated with COVID-19 have been reported, making COVID-19 a major health emergency.

Antiviral drugs that are being evaluated as potential treatments for COVID-19 include lopinavir/ritonavir (LPV/RTV; used in the treatment of HIV infection) and remdesivir (RDV, GS-5734<sup>TM</sup>). In a study of Severe Acute Respiratory Syndrome (SARS), a significant reduction in acute respiratory distress syndrome/mortality was observed in 41 patients treated with the combination of LPV/RTV, compared with 111 patients receiving monotherapy ribavirin (2.4 % vs 28.8%, p 0.001). However, the use of historical control data does not allow for a reliable estimation of efficacy. Additionally, LPV/RTV has multiple known adverse reactions such as prolonged QT interval, severe gastrointestinal reactions, abnormal blood glucose, pancreatitis, hepatic impairment, and elevated blood lipids. It has multiple drug-to-drug interactions with many commonly used drugs in clinical practice; thus, its clinical safety is not determined. Remdesivir shows potent in vitro activity against the human pathogenic CoVs Middle East Respiratory Syndrome (MERS)-CoV and SARS-CoV in multiple relevant human cell types. In a mouse model of MERS-CoV infection, both prophylactic and therapeutic RDV significantly improved pulmonary function and reduce lung viral loads and severe lung pathology compared with vehicle control animals. In contrast, prophylactic LPV/RTV + interferon-beta (LPV/RTV-IFNb) slightly reduced viral loads without impacting other disease parameters. Therapeutic LPV/RTV-IFNb improves pulmonary function but did not reduce virus replication or severe lung pathology {Sheahan 2020}.

The evaluation of the safety and potential efficacy of RDV in people with COVID-19 is urgently needed.

# **1.2.** Remdesivir (RDV, GS-5734)

Remdesivir is being developed by Gilead Sciences, Inc. (Gilead) and is formulated for intravenous (IV) administration.

### 1.2.1. General Information

Remdesivir is a nucleotide prodrug that is intracellularly metabolized into an analog of adenosine triphosphate that inhibits viral RNA polymerases and has broad spectrum activity against members of the filoviruses (eg, Ebola virus [EBOV], Marburg virus [MARV]), CoVs (eg, SARS-CoV, MERS-CoV), and paramyxoviruses (eg, respiratory syncytial virus [RSV], Nipah virus, and Hendra virus). For further information on RDV, refer to the current investigator's brochure (IB) for RDV. Information in the IB includes:

- Nonclinical pharmacokinetic (PK) and in vitro metabolism
- Nonclinical pharmacology and toxicology
- Clinical experience

Additional relevant information regarding RDV are described below.

# 1.2.2. Preclinical Pharmacology and Toxicology

Recent results from initial in vitro testing performed at the China CDC in collaboration with Gilead showed that RDV has potent antiviral activity against SARS-CoV-2 in Vero cells (EC50 0.137  $\mu$ M). In another study conducted by the Wuhan Institute of Virology, RDV also showed in vitro activity against SARS-CoV-2 in Vero cells (EC50 0.77  $\mu$ M) {Wang 2020}. Gilead notes that the study from the Wuhan Institute of Virology was conducted externally with drug not supplied by Gilead. Researchers in the United States (US) and China are continuing to test RDV against clinical isolates of SARS-CoV-2 using drug supplied by Gilead in multiple relevant cell types that are known to more efficiently metabolize RDV into its active triphosphate form compared with Vero cells.

### 1.3. Rationale for This Study

There is currently no approved treatment available for COVID-19 infection. The recommendation for using RDV as treatment of COVID-19 is based on the in vitro and in vivo activity of RDV against SARS-CoV-2 and other highly pathogenic human CoVs, MERS-CoV and SARS-CoV.

Remdesivir has acceptable nonclinical tolerability and safety profiles and exhibits in vivo prophylactic and therapeutic efficacy against SARS-CoV and MERS-CoV infection in mice and MERS-CoV infection in rhesus monkeys. In addition, RDV has been shown to be safe and tolerable; with a safety database of over 500 individuals who have received RDV to date. Key attributes of the RDV nonclinical and clinical profile supporting its use for treatment of COVID-19 are as follows:

 Initial in vitro testing performed at the China CDC in collaboration with Gilead showed that RDV has potent antiviral activity against SARS-CoV-2 in Vero cells (EC<sub>50</sub> 0.137 μM).
 Remdesivir has also shown potent in vitro activity against the human pathogenic CoVs MERS-CoV and SARS-CoV in multiple relevant human cell types.

- The PK profile of RDV in nonhuman primates (NHPs) and other relevant animal species indicates high and persistent levels of pharmacologically active nucleoside triphosphate metabolite in peripheral blood mononuclear cells (PBMCs), supporting once daily IV administration as a 30-minute infusion.
- Remdesivir demonstrated prophylactic and therapeutic efficacy in a mouse model of SARS- CoV pathogenesis. Administration of 25 mg/kg RDV subcutaneously twice daily beginning 1 day before or 1 day after SARS-CoV inoculation resulted in significantly reduced lung viral load and improved clinical signs of disease as well as lung function {Sheahan 2017}.
- In a mouse model of MERS-CoV pathogenesis, both prophylactic and therapeutic administration of 25 mg/kg RDV subcutaneously twice daily improved pulmonary function and reduced lung viral loads and severe lung pathology. In contrast, prophylactic LPV/RTV IFNb slightly reduced viral loads without impacting other disease parameters. Therapeutic LPV/RTV-IFNb improved pulmonary function but did not reduce virus replication or severe lung pathology {Sheahan 2020}.
- Remdesivir also showed prophylactic and therapeutic efficacy in MERS-CoV-infected rhesus monkeys of Indian origin. Administration of RDV at 10 mg/kg (see RDV IB) or 5 mg/kg once daily for 7 days using IV bolus injection beginning 1 day prior to MERS-CoV inoculation resulted in a significant reduction of clinical scores, clinical signs of respiratory disease, and viral RNA levels compared to vehicle-treated animals. Therapeutic RDV treatment of 5 mg/kg once daily using IV bolus injection initiated 12 hours post-inoculation also resulted in reduced clinical signs, reduced virus replication in the lungs, and decreased presence and severity of lung lesions {De Wit 2020}.

Remdesivir has a favorable clinical safety profile based on approximately 500 individuals who received RDV primarily as healthy volunteers in Phase 1 studies and individuals with acute EBOV infection.

The design of enrollment in two parts will allow the selection of a preferred duration of treatment to be determined and then allow continued access to RDV and data collection for eligible participants. In addition, further safety data will be obtained.

#### 1.4. Rationale for Dose Selection of Remdesivir

The proposed regimen for the treatment of established CoV infection, including SARS-CoV and MERS-CoV, is as follows: single RDV 200 mg IV loading dose on Day 1 of treatment followed by 100 mg IV once-daily maintenance doses for a total of up to 10 days of dosing. The proposed dosing regimen is based on efficacy studies in MERS-infected rhesus monkeys treated with RDV (Studies PC-399-2037 and PC-399-2038) and based on clinical safety data in approximately 500 patients including healthy volunteers and individuals with acute EBOV infection.

In the nonclinical studies, RDV was administered at 10 mg/kg (Study PC-399-2038) or 5 mg/kg (Study PC-399-2037) once daily for 7 days using IV bolus injection beginning either 1 day prior to or 12 hours after (5 mg/kg only) MERS-CoV inoculation. Remdesivir treatment was

efficacious at reducing viral titers in the lung and alleviating clinical disease signs (RDV IB; {De Wit 2020}). Toxicology studies in cynomolgus monkeys and rats and safety and PK studies in healthy volunteers support the safety of the proposed dose. Overall, RDV has a favorable PK and safety profile that supports evaluation of a 200 mg loading and a 100 mg daily dose that has potential to be efficacious in adult patients with COVID-19.

The optimal duration of therapy with RDV remains unknown. However, other agents for acute antiviral infection, for example oseltamivir phosphate {TAMIFLU® 2019}, have treatment courses ranging from 5 days duration. There is considerable potential patient benefit and societal benefit in identifying the minimum duration that will be effective.

## 1.4.1. Pediatric Dosing

As with adult dose, the efficacious dose of RDV against SARS-CoV-2 remains to be established.

Dose selection of remdesivir (RDV) in EBOV infected pediatric patients was informed by a physiologically-based pharmacokinetic (PBPK) model implemented in SimCYP (v.17, Certara). Briefly, a PBPK model was developed to characterize the PK of RDV and the primary circulating nucleoside metabolite, GS-441524, in adults. The model was verified based on its ability to describe the mean and variability of the adult exposures using data from the RDV Phase 1 program (GS-US-399-1812). The adult PBPK model was subsequently used to simulate steady-state pediatric (age range 0 to 18 years) exposures (AUC<sub>tau</sub>), accounting for age-dependent changes in organ volume/size (liver and kidney), esterase expression, plasma protein binding, and organ blood flow.

These simulations do not account for diminished liver or kidney function due to SARS-CoV-2 infection and/or COVID-19 progression because the impact of infection/disease progression on the PK of remdesivir and GS-441524 is currently unknown.

The results of these simulations indicate:

For pediatric patients with body weight  $\geq$  40 kg, a 200 mg loading dose followed by 100 mg once-daily maintenance doses of remdesivir (ie, the adult dosage regimen) should be administered. Use of the adult dose in these pediatric patients is expected to maintain exposures of both remdesivir and GS-441524 generally within those expected at the therapeutic doses and which were previously observed to be well tolerated in healthy volunteers.

### 1.5. Risk/Benefit Assessment for the Study

Potential risks associated with the study include unknown adverse events (AEs) and laboratory abnormalities. Although not specifically evaluated yet, adolescents with COVID-19 who receive RDV are expected to have a similar safety profile as adults; no additional safety monitoring is required for adolescent participants and no dose adjustments are required. No differing safety profile has been reported for the adolescents with EBOV who received RDV in clinical trials. Accordingly, the risk:benefit profile, described below, is the same for adolescents and adults.

A pertinent specific risk for participants in this study is the potential for transient, Grade  $\leq 2$ , treatment-emergent elevations in alanine aminotransferase (ALT) and aspartate aminotransferase (AST), which were observed after multiple daily RDV administrations in Studies GS-US-399-1954 and GS-US-399-5505.

To date in human studies, no serious adverse events (SAEs) have occurred in healthy individuals who have received at least 1 dose of RDV. Remdesivir has been tested in healthy volunteers as a single ascending dose over a dose range of 3 to 225 mg and in a multi-dose study of 150 mg for up to 14 days and at 200 mg loading dose followed by 100 mg for a total of 10 days.

In nonclinical animal studies, toxicity findings were consistent with dose-dependent and reversible kidney injury and dysfunction. The clinical significance of the nephrotoxicity noted in animal species is unknown. The etiology of reversible kidney injury observed in rats is consistent with the ability of rat renal organic anion transporters (OATs), but not human OATs, to efficiently interact with blood metabolites of RDV, particularly GS-704277. This effect may lead to proportionally higher intracellular accumulation of drug metabolites in renal rat tubules, leading to kidney injury.

The 200 mg loading dose with 8 g of sulfobutylether  $\beta$ -cyclodextrin sodium (SBECD) on Day 1 will be followed by 100 mg of RDV each day for 4 or 9 days with 4 g of SBECD, which is within the range of daily SBECD administration considered safe in humans. A total of 250 mg/kg/day of SBECD is considered safe by the European Medicines Agency and is therefore safe for people with weight over 32 kg. The 100 mg dose prepared in 0.9% saline will be hypertonic relative to human serum osmolality but approaches the normal physiological osmolar range for humans. The RDV regimen consisting of a loading dose of 200 mg followed by RDV 100 mg daily for up to 9 days is not anticipated to pose a safety risk to participants enrolled in this study.

There are currently no data available on the interaction of RDV and other investigational agents. Administering RDV concurrent with other investigational anti-CoV agents may lead to antagonism or synergy or have no effect.

The risk mitigation strategy for this study includes restriction of the study population to those without a history of significant renal or hepatic disease:

- Exclusion of participants with ALT  $> 5 \times ULN$
- Exclusion of participants with an estimated glomerular filtration rate (eGFR) < 50 mL/min
- Exclusion of coadministration of other investigational agents against COVID-19
- Serum chemistry assessments, including liver function testing, will be closely monitored during the study period.

There are currently no investigational agents with demonstrated clinical efficacy or approved treatments for COVID-19. The timely evaluation of a safe and effective antiviral agent that works by directly and selectively blocking the virus replication and is broadly efficacious against COVID-19 addresses a serious unmet medical need. In consideration of the information included in this protocol, the overall risks to participants are outweighed by the potential benefits of RDV experimental therapy for the treatment of COVID-19. The benefit-risk balance for this study is considered positive.

# 1.6. Compliance

This study will be conducted in compliance with this protocol, Good Clinical Practice (GCP), and all applicable regulatory requirements.

# 2. OBJECTIVES

The purpose of this study is to provide RDV to participants with severe COVID-19.

The primary objective of this study is as follows:

• To evaluate the efficacy of 2 RDV regimens with respect to clinical status assessed by a 7-point ordinal scale on Day 14

The secondary objective of this study is as follows:

• To evaluate the safety and tolerability of RDV

### 3. STUDY DESIGN

Part A of this study is a randomized, open-label, multicenter study of RDV in participants with severe COVID-19 infection. Part B is a two treatment group multicenter study of RDV in participants with severe COVID-19 infection. Treatment group assignment is based on whether the participant is on mechanical ventilation at treatment assignment. All participants will continue to receive SOC therapy according to local guidelines.

# 3.1. Endpoints

The primary endpoint of this study is:

• Clinical status assessed by a 7-point ordinal scale on Day 14

The secondary endpoint of this study is:

• The proportion of participants with treatment emergent AEs

Other endpoints of interest are:

- Time to  $SpO_2 > 94\%$  on room air
- Time to first negative SARS-CoV-2 polymerase chain reaction (PCR)
- Duration of oxygen therapy (days)
- Duration of hospitalization (days)
- All cause mortality at Day 28
- Time to clinical improvement (days): Clinical improvement is defined as a  $\geq$  2-point improvement from Day 1 on a 7-point ordinal scale

### CCI

• The proportion of participants in the Mechanically Ventilated Treatment Group and Extension Treatment Group with treatment-emergent AEs

### 3.2. Study Design

Part A of this study is a randomized, open-label, multicenter study of RDV in participants with severe COVID-19 infection. Eligible participants will be randomized in equal proportions to 1 of 2 treatment groups. No stratification will be performed. Part B is a two treatment group multicenter study of RDV in participants with severe COVID-19 infection.

# 3.3. Study Treatments

In Part A, approximately 400 participants who meet all eligibility criteria and who are not mechanically ventilated may be randomized in a 1:1 ratio into 1 of the following treatment groups:

**Treatment Group 1:** continued standard of care therapy together with IV RDV 200 mg on Day 1 followed by IV RDV 100 mg on Days 2, 3, 4, and 5

**Treatment Group 2:** continued standard of care therapy together with IV RDV 200 mg on Day 1 followed by IV RDV 100 mg on Days 2, 3, 4, 5, 6, 7, 8, 9, and 10

In Part B, an additional approximately 5600 participants who meet all of the eligibility criteria may receive:

**Mechanically Ventilated Treatment Group:** continued standard of care therapy together with IV RDV 200 mg on Day 1 followed by IV RDV 100 mg on Days 2, 3, 4, 5, 6, 7, 8, 9, and 10

**Extension Treatment Group:** continued standard of care therapy together with IV RDV 200 mg on Day 1 followed by IV RDV 100 mg on Days 2, 3, 4, 5, 6, 7, 8, 9, and 10 unless the 5-day dosing regimen used in Treatment Group 1 of Part A is selected. If treatment for 5 days is selected, all participants in the Extension Treatment Group and all new participants will be reassigned to receive treatment for a total of 5 days. National and local regulatory authorities will be informed.

Participants in Part A of the study will be the primary efficacy population. Participants enrolled in Part B will have data reported descriptively at study completion.

### 3.4. **Duration of Treatment**

Participants will receive study treatment with RDV for 5 days (Treatment Group 1), 10 days (Treatment Group 2), 10 days (Mechanically Ventilated Treatment Group), or either 5 or 10 days (Extension Treatment Group). If the participant is discharged, RDV treatment will stop at that time.

### 3.5. Discontinuation Criteria

Study drug dosing in an individual subject will be placed on hold and may be discontinued, following a review of all available clinical data by the medical monitor and discussion with the investigator, if any of the following occurs:

- Any SAE or  $\geq$  Grade 3 AE suspected to be related to RDV.
- Any elevations in ALT  $> 5 \times$  ULN; or ALT  $> 3 \times$  ULN and total bilirubin  $> 2 \times$ ULN, confirmed by immediate repeat testing.
- Creatinine clearance < 30mL/min

Discontinuation of study medication is not a seriousness criterion.

# 3.6. End of Study

The end of the study will be the last participant's last observation (or visit).

# 3.7. Post Study Care

The long-term care of the participant will remain the responsibility of their primary treating physician. Remdesivir is being supplied with curative intent. There is no provision for post-study availability.

## 4. SUBJECT POPULATION

### 4.1. Number of Subjects and Subject Selection

In Part A, approximately 400 participants will be randomized in a 1:1 ratio into 1 of 2 treatment groups. In Part B, up to approximately 5600 participants may be assigned to 1 of 2 treatment groups. Rescreening may occur at the investigator's discretion.

### 4.1.1. Subject Replacement

Subjects who discontinue prior to the end of study will not be replaced.

#### 4.2. Inclusion Criteria

Subjects must meet all of the following inclusion criteria to be eligible for participation in this study:

- 1) Willing and able to provide written informed consent, or with a legal representative who can provide informed consent, or enrolled under ICH E6(R2) 4.8.15 emergency use provisions as deemed necessary by the investigator (participants ≥ 18 years of age), or willing and able to provide assent (participants ≥ 12 and < 18 years of age, where locally and nationally approved) prior to performing study procedures. For participants ≥ 12 and < 18 years of age, a parent or legal guardian willing and able to provide written informed consent prior to performing study procedures
- 2) Aged  $\geq$  18 years (at all sites), or aged  $\geq$  12 and < 18 years of age weighing  $\geq$  40 kg (where permitted according to local law and approved nationally and by the relevant institutional review board [IRB] or independent ethics committee [IEC])
- 3) SARS-CoV-2 infection confirmed by PCR test ≤ 4 days before randomization
- 4) Currently hospitalized
- 5) SpO<sub>2</sub>  $\leq$  94% on room air or requiring supplemental oxygen at screening
- 6) Radiographic evidence of pulmonary infiltrates
- 7) Men and women of childbearing potential who engage in heterosexual intercourse must agree to use protocol specified method(s) of contraception as described in Appendix 3.

# 4.3. Exclusion Criteria

Subjects who meet *any* of the following exclusion criteria are not to be enrolled in this study:

- 1) Participation in any other clinical trial of an experimental treatment for COVID-19
- 2) Concurrent treatment with other agents with actual or possible direct acting antiviral activity against SARS-CoV-2 < 24 hours prior to study drug dosing
- 3) Evidence of multiorgan failure
- 4) Mechanically ventilated (including V-V ECMO) ≥ 5 days, or any duration of V-A ECMO
- 5) ALT or AST  $> 5 \times ULN$
- 6) Creatinine clearance < 50 mL/min using the Cockcroft-Gault formula for participants ≥ 18 years of age {Cockcroft 1976} and Schwartz Formula for participants < 18 years of age
- 7) Positive pregnancy test (Appendix 3)
- 8) Breastfeeding woman
- 9) Known hypersensitivity to the study drug, the metabolites, or formulation excipient

### 5. INVESTIGATIONAL MEDICINAL PRODUCTS

### 5.1. Randomization, Blinding, and Treatment Codes Access

### 5.1.1. Randomization

Subjects who meet eligibility criteria will be randomized in a 1:1 ratio to 1 of 2 treatment groups on Day 1 using an IWRS and assigned a subject number. Randomization will not be stratified.

# 5.1.2. Blinding

Blinding of treatment assignments or data will not be performed in this study.

### 5.2. Description and Handling of Remdesivir

### **5.2.1.** Formulation

Remdesivir for injection, 100 mg, is a preservative-free, white to off-white to yellow, lyophilized solid containing 100 mg of GS-5734 that is to be reconstituted with sterile water for injection and diluted into 0.9% saline prior to administration by IV infusion.

In addition to the active ingredient, RDV for injection, 100 mg, contains the following inactive ingredients: betadex sulfobutyl ether sodium (SBECD), water for injection, hydrochloric acid, and sodium hydroxide. Hydrochloric acid and sodium hydroxide are used to adjust the formulation to a pH of 3.0 to 4.0.

### 5.2.2. Packaging and Labeling

Remdesivir for injection, 100 mg, is supplied as a sterile product in a single-use, 30 mL Type I clear glass vial. Each vial is sealed with a fluoro-resin laminated rubber stopper and an aluminum overseal with a red, plastic flip-off cap.

Remdesivir for injection, 100 mg, shall be labeled to meet all applicable requirements of the US Food and Drug Administration (FDA), EU Guideline to Good Manufacturing Practice - Annex 13 (Investigational Medicinal Products), the J-GCP (Ministerial Ordinance on Good Clinical Practice for Drugs), as applicable, and/or other local regulations.

# 5.2.3. Storage and Handling

Remdesivir for injection, 100 mg, should be stored below 30 °C (86 °F) prior to use. Storage conditions are specified on the label. Until dispensed for dosing, all vials of study drugs should be stored in a securely locked area, accessible only to authorized site personnel.

To ensure the sterility, stability, and proper identification, study drug(s) should not be stored in a container other than the container in which they were supplied.

Measures that minimize drug contact with the body should always be considered during handling, preparation, and disposal procedures.

Remdesivir for injection, 100 mg, is recommended to be reconstituted and diluted on the same day as administration. Remdesivir for injection, 100 mg, does not contain any preservative and is intended for single-use. Any unused RDV material should be discarded.

### 5.3. Dosage and Administration of Remdesivir

Remdesivir for injection, 100 mg, will be provided by Gilead. In Part A, participants in Treatment Groups 1 and 2 will receive RDV 200 mg on Day 1 followed by IV RDV 100 mg on Days 2, 3, 4, and 5. Participants in Treatment Group 2 will also receive RDV 100 mg on Days 6, 7, 8, 9, and 10. In Part B, participants in the Mechanically Ventilated Treatment Group will receive IV RDV 200 mg on Day 1 followed by IV RDV 100 mg on Days 2, 3, 4, 5, 6, 7, 8, 9, and 10. Participants in the Extension Treatment Group will also receive IV RDV 200 mg on Day 1 followed by IV RDV 100 mg on Days 2, 3, 4, 5, 6, 7, 8, 9, and 10 unless the 5-day dosing regimen used in Treatment Group 1 of Part A is selected. If treatment for 5 days is selected, all participants in the Extension Treatment Group and all new participants will be reassigned to receive treatment for a total of 5 days. Remdesivir treatment will be stopped at discharge regardless of the scheduled duration of therapy. Remdesivir will be administered over 30 minutes where possible.

# 5.4. Accountability for Investigational Medicinal Product

The investigator is responsible for ensuring adequate accountability of all used and unused study drug. This includes acknowledgment of receipt of each shipment of study drug (quantity and condition).

Each study site must keep accountability records that capture:

- The date received and quantity of study drug kits
- The date, subject number, and the study drug kit number dispensed
- The date, quantity of used and unused study drug returned, along with the initials of the person recording the information

# 5.4.1. Investigational Medicinal Product Return or Disposal

Gilead recommends that used and unused study drug supplies be destroyed at the site. If the site has an appropriate SOP for drug destruction as determined by Gilead, the site may destroy used (empty or partially empty) and unused study drug supplies in accordance with that site's approved SOP. A copy of the site's approved SOP will be obtained for eTMF. If study drug is destroyed on site, the investigator must maintain accurate records for all study drugs destroyed. Records must show the identification and quantity of each unit destroyed, the method of destruction, and the person who disposed of the study drug. Upon study completion, copies of the study drug accountability records must be filed at the site. Another copy will be returned to Gilead.

If the site does not have an appropriate SOP for drug destruction, used and unused study drug supplies are to be sent to the designated disposal facility for destruction. The study monitor will provide instructions for return.

The study monitor will review study drug supplies and associated records at periodic intervals.

For both disposal options listed above, the study monitor must first perform drug accountability during an on-site monitoring visit.

#### 5.5. Prior and Concomitant Medications

Concomitant use of the following is prohibited in participants receiving RDV:

- Traditional herbal treatments including herb sho-saiko-to (or Xiao-Shai-Hu-Tang)
- Investigational agents with putative antiviral activity for COVID-19 including approved HIV protease inhibitors such as lopinavir/ritonavir, chloroquine, interferon, etc.

Concomitant use of investigational agents such as approved HIV protease inhibitors like lopinavir/ritonavir, chloroquine, etc while receiving RDV is prohibited due to lack of evidence on additive or synergistic effects and potential for an increased risk of transaminase elevations.

Medications will be assessed only from Day 1 prior to enrollment to Day 14 or discharge, whichever is earlier.

### 6. STUDY PROCEDURES

The study procedures to be conducted for each subject enrolled in the study are presented in tabular form in Appendix 2 and described in the text that follows.

The investigator must document any deviation from the protocol procedures and notify the Gilead or contract research organization (CRO).

### 6.1. Subject Enrollment and Treatment Assignment

Entry into screening does not guarantee enrollment into the study. In order to manage the total study enrollment, Gilead, at its sole discretion, may suspend screening and/or enrollment at any site or study-wide at any time.

#### 6.2. Pretreatment Assessments

# 6.2.1. Screening Visit

Subjects will be screened within 2 days before randomization and dosing to determine eligibility for participation in the study.

Obtain written informed consent, or with a legal representative who can provide informed consent, or enrolled under ICH E6(R2) 4.8.15 emergency use provisions as deemed necessary by the investigator (participants  $\geq$  18 years of age), or obtain assent (participants age  $\geq$ 12 to <18, where locally and nationally approved)

After the informed consent the following assessments are performed to determine eligibility requirements as specified in the inclusion and exclusion criteria:

- Focused medical history including the following information (eg, date of first symptoms, overall symptoms, exposure source, demographics, baseline characteristics), allergies and medical history
- Review and record medications and therapies for this current illness
- Counsel subjects to use adequate birth control methods required during the trial to avoid pregnancy
- Targeted physical examination including, vital signs (heart rate, temperature, blood pressure), body weight, and height
- Documentation of respiratory status:

Respiratory Rate

Oxygen supplementation: room air, low flow O<sub>2</sub> (L/min and %), high flow O<sub>2</sub> (L/min and %), CPAP/BIPAP (FiO<sub>2</sub> or %), mechanical ventilation (FiO<sub>2</sub> or %), ECMO

Oxygenation: SpO<sub>2</sub> or PaO<sub>2</sub>

Radiographic findings

- Obtain blood samples if not done in the preceding 48 hours for creatinine, creatinine clearance, ALT and AST
- Pregnancy test (for women of childbearing potential)
- Record any SAEs and all AEs related to protocol-mandated procedures occurring after signing of the consent (or assent) form.

Study subjects who qualify should be immediately randomized. Randomization and dosing should occur on the same day if possible.

# 6.2.2. Baseline/Day 1 Assessments

The following evaluations are to be completed at the Day 1 visit. The investigator must have confirmed eligibility before proceeding with randomization (Part A) or treatment assignment (Part B) on the Day 1 visit. If the screening and Day 1 visits occur within one day, no procedures need to be repeated. Participants must complete the following assessments before being administered study drug:

- Physical examination including vital signs (heart rate, temperature, blood pressure, and body weight)
- Documentation of respiratory status:

Respiratory rate

Oxygen supplementation: room air, low flow O<sub>2</sub> (L/min and %), high flow O<sub>2</sub> (L/min and %), CPAP/BIPAP (FiO<sub>2</sub> or %), mechanical ventilation (FiO<sub>2</sub> or %), ECMO

Oxygenation: SpO<sub>2</sub> or PaO<sub>2</sub>

Radiographic findings (if available)

- Review AEs and document concomitant medications
- Obtain blood samples for white blood cell count, hemoglobin and/or hematocrit, platelets, creatinine and creatinine clearance, glucose, total bilirubin, ALT, AST
- Review the Ordinal Scale (see Section 6.9)

# 6.3. Daily Study Assessments (Days 2-14)

The following evaluations are to be completed daily from Days 2 14 or until discharge whichever comes earlier:

- Vital signs (heart rate, temperature, blood pressure), body weight (if available).
- A symptom-directed (targeted) physical examination will be performed to evaluate for any possible adverse event
- Documentation of respiratory status:

Respiratory rate

Oxygen supplementation: room air, low flow O<sub>2</sub> (L/min and %), high flow O<sub>2</sub> (L/min and %), CPAP/BIPAP (FiO<sub>2</sub> or %), mechanical ventilation (FiO<sub>2</sub> or %), ECMO

Oxygenation: SpO<sub>2</sub> or PaO<sub>2</sub>

Radiographic findings (if available)

- SARS-CoV-2 testing results if available should be reported
- Review of AEs and document concomitant medications
- Review Ordinal Scale (Section 6.9)

# 6.4. Additional Assessments

The following evaluations are to be completed at the following visits or until discharge, whichever comes earlier:

 Safety laboratory tests (white blood cell count, hemoglobin and/or hematocrit, platelets, creatinine and creatinine clearance, glucose, total bilirubin, ALT, AST) are to be completed at Days 3, 5, 8, 10, and 14

# 6.5. Day 28 Follow up Assessment (±5 Days)

The following evaluations are to be completed if this visit is conducted in person. For participants who have been discharged from hospital, the final evaluation can be made by phone. Only AE and concomitant medication and ordinal scale (if discharged on or after Day 14) review are to be completed if visit is conducted by phone.

• Physical examination and vital signs (heart rate, temperature, blood pressure)

• Documentation of respiratory status:

Respiratory rate

— Oxygen supplementation: room air, low flow O<sub>2</sub> (L/min and %), high flow O<sub>2</sub> (L/min and %), CPAP/BIPAP (FiO<sub>2</sub> or %), mechanical ventilation (FiO<sub>2</sub> or %), ECMO

Oxygenation: SpO<sub>2</sub> or PaO<sub>2</sub>

Radiographic findings (if available)

- Review AEs and document concomitant medications
- Review the Ordinal Scale (Section 6.9). If subject was not discharged by Day 14, any change in category and the date of any change in category from Day 14 to discharge (or Day 28) should be recorded

### 6.6. Clinical Laboratory Assessments

Clinical laboratory assessments are required at screening, Days 1, 3, 5, 8, 10 and 14 or until discharge whichever comes earlier. Clinical laboratory assessments at other days may be conducted if required by clinical need or local practice. All laboratory testing will be completed by local laboratories. From Day 1 to Day 14, at specified timepoints, the sponsor will be provided with results for the following analytes: white blood cell count, hemoglobin and/or hematocrit, platelets, creatinine and creatinine clearance, glucose, total bilirubin, ALT, AST, and any SARS-CoV-2 testing.

SARS-CoV-2 testing may include RT-qPCR to detect or quantify SARS-CoV-2 or virus sequencing results. If feasible, oropharyngeal, saliva, sputum, stool, and/or blood samples may be collected and assayed using RT-qPCR to quantify SARS-CoV-2 viral load. Pretreatment and posttreatment samples with detectable SARS-CoV-2 may be sequenced for resistance monitoring of the viral polymerase gene if possible.

For all clinical laboratory tests at Day 1, at least the most recent result before dosing should be used. For other tests, preferably enter all results if the most recent result before dosing is not available. When more than 1 result is available in a calendar day, at minimum, results should be reported as indicated in Table 1. All SARS-CoV-2 results should be provided.

Table 1. Data Entry Requirements When Only One Result of Multiple Results Is Recorded for a Given Day

| Test Name | Minimum Data to be Recorded Highest result |
|---|---|
| Alanine aminotransferase | |
| Aspartate aminotransferase | Highest result |
| Creatinine | Highest result |
| Glucose | Lowest result (hypoglycemia) Highest result (hyperglycemia) if outside normal range |
| Total bilirubin | Highest result |
| Hematocrit | Lowest result |
| Hemoglobin | Lowest result |
| Platelets | Lowest result |
| White Blood Cells | Lowest result |
| Creatinine Clearance (Cockcroft-Gault or Schwarz preferred) | Lowest result |

# 6.7. Physical Examination

A targeted physical examination and vital signs (heart rate, respiratory rate, temperature, blood pressure, SpO<sub>2</sub> or PaO<sub>2</sub>) should be performed at least daily.



# 6.9. Ordinal Scale

The ordinal scale is an assessment of the clinical status at a given study day. Each day, the worst (i.e. lowest ordinal) score from the previous day will be recorded. i.e. on Day 3, the lowest ordinal score from Day 2 is obtained and recorded for Day 2. The scale is as follows:

- 1. Death
- 2. Hospitalized, on invasive mechanical ventilation or ECMO
- 3. Hospitalized, on non-invasive ventilation or high flow oxygen devices

- 4. Hospitalized, requiring low flow supplemental oxygen
- 5. Hospitalized, not requiring supplemental oxygen requiring ongoing medical care (COVID-19 related or otherwise)
- 6. Hospitalized, not requiring supplemental oxygen no longer requires ongoing medical care (other than per protocol RDV administration)
- 7. Not hospitalized

### **6.10.** Post-treatment Assessments

No assessments are required after Day 28.

### 6.11. Assessments for Early Discontinuation from Study

If a subject discontinues study dosing (for example, as a result of an AE or clinically significant laboratory abnormality), every attempt should be made to keep the subject in the study and continue to perform the required study-related follow-up and procedures (see Section 3.5, Discontinuation Criteria). If this is not possible or acceptable to the subject or investigator, the subject may be withdrawn from the study.

# 6.11.1. Criteria for Discontinuation of Study Treatment

Study medication may be discontinued in the following instances:

- Discharge from the hospital/institution
- Intercurrent illness that would, in the judgment of the investigator, affect assessments of clinical status to a significant degree. Following resolution of intercurrent illness, the subject may resume study dosing at the discretion of the investigator.
- Unacceptable toxicity, or toxicity that, in the judgment of the investigator, compromises the ability to continue study-specific procedures or is considered to not be in the subject's best interest
- Subject request to discontinue for any reason
- Subject noncompliance
- Pregnancy during the study; refer to Appendix 3
- Discontinuation of the study at the request of Gilead, a regulatory agency or an IRB or IEC

# 6.12. End of Study

The end of the study will occur when the last participant's last observation (or visit).

# 6.13. Post Study Care

The long-term care of the participant will remain the responsibility of their primary treating physician. Remdesivir is being supplied with curative intent. There is no provision for post-study availability.

# 6.14. Sample Disposition and Storage (Non-PK Samples)

Samples will be processed and retained according to local practice and the regulations pertaining to each institution. No samples will be obtained or retained by Gilead.



## 7. ADVERSE EVENTS AND TOXICITY MANAGEMENT

#### 7.1. Definitions of Adverse Events and Serious Adverse Events

#### 7.1.1. Adverse Events

An AE is any untoward medical occurrence in a clinical study subject administered an investigational product, which does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and/or unintended sign, symptom, or disease temporally associated with the use of an investigational product, whether or not considered related to the investigational product. AEs may also include pretreatment or posttreatment complications that occur as a result of protocol specified procedures or special situations (Section 7.6).

An AE does not include the following:

- Medical or surgical procedures such as surgery, endoscopy, tooth extraction, and transfusion. The condition that led to the procedure may be an AE and must be reported.
- Preexisting diseases, conditions, or laboratory abnormalities present or detected before the screening visit that do not worsen
- Situations where an untoward medical occurrence has not occurred (eg, hospitalization for elective surgery, social and/or convenience admissions)
- Overdose without clinical sequelae (Section 7.6.1)
- Any medical condition or clinically significant laboratory abnormality with an onset date before the consent form is signed and not related to a protocol-associated procedure is not an AE. It is considered to be preexisting and should be documented as medical history.

Preexisting events or conditions that increase in severity or change in nature after the consent form is signed or as a consequence of participation in the clinical study will be considered AEs

## 7.1.2. Serious Adverse Events

A SAE is defined as an event that, at any dose, results in the following:

- Death
- Life-threatening (Note: The term "life-threatening" in the definition of "serious" refers to an event in which the subject was at risk of death at the time of the event; it does not refer to an event that hypothetically might have caused death if it were more severe.)
- In-patient hospitalization or prolongation of existing hospitalization
- Persistent or significant disability/incapacity
- A congenital anomaly/birth defect

• A medically important event or reaction: such events may not be immediately life-threatening or result in death or hospitalization but may jeopardize the subject or may require intervention to prevent one of the other outcomes constituting SAEs. Medical and scientific judgment must be exercised to determine whether such an event is a reportable under expedited reporting rules. Examples of medically important events include intensive treatment in an emergency room or at home for allergic bronchospasm; blood dyscrasias or convulsions that do not result in hospitalization; and development of drug dependency or drug abuse.

### 7.2. Assessment of Adverse Events and Serious Adverse Events

The investigator or qualified subinvestigator is responsible for assessing AEs and SAEs for causality and severity, and for final review and confirmation of accuracy of event information and assessments.

## 7.2.1. Assessment of Causality for Study Drugs and Procedures

The investigator or qualified subinvestigator is responsible for assessing the relationship to study drug using clinical judgment and the following considerations:

- No: Evidence exists that the AE has an etiology other than the study drug. For SAEs, an alternative causality must be provided (eg, preexisting condition, underlying disease, intercurrent illness, or concomitant medication).
- Yes: There is reasonable possibility that the AE may have been caused by the study drug.

It should be emphasized that ineffective treatment should not be considered as causally related in the context of AE reporting.

The relationship to study procedures (eg, invasive procedures such as venipuncture or biopsy) should be assessed using the following considerations:

- No: Evidence exists that the AE has an etiology other than the study procedure.
- Yes: The AE occurred as a result of protocol procedures (eg, venipuncture)

### 7.2.2. Assessment of Severity

The severity of AEs will be graded using the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 dated July 2017. For each episode, the highest grade attained should be reported as defined in the grading scale. The DAIDS scale is available at the following location:

https://rsc.niaid.nih.gov/sites/default/files/daidsgradingcorrectedv21.pdf
# 7.3. Investigator Requirements and Instructions for Reporting Adverse Events and Serious Adverse Events

## 7.3.1. Requirements for Collection Prior to Study Drug Initiation

After informed consent, but prior to initiation of study medication, the following types of events must be reported on the applicable eCRFs: all SAEs and AE related to protocol-mandated procedures.

#### 7.3.2. Adverse Events

Following initiation of study medication, collect all AEs, regardless of cause or relationship, throughout the duration of the study, including the protocol-required post treatment follow-up period must be reported on the eCRFs as instructed.

All AEs and clinically significant laboratory abnormalities should be followed up until resolution or stability of the abnormality has been demonstrated, if possible. Gilead may request that certain AEs be followed beyond the protocol-defined follow-up period.

#### 7.3.3. Serious Adverse Events

All SAEs, regardless of cause or relationship, that occurs after the subject first consents to participate in the study (ie, signing the informed consent) and throughout the duration of the study, including the protocol-required post treatment follow-up period must be reported on the applicable eCRFs and Pharmacovigilance an Epidemiology (PVE) as instructed below in this section. This also includes any SAEs resulting from protocol-associated procedures performed after informed consent is signed.

Any SAEs and deaths that occur after the post-treatment follow-up visit but within 30-days of the last dose of study drug, regardless of causality, should also be reported.

Investigators are not obligated to actively seek SAEs after the protocol-defined follow-up period; however, if the investigator learns of any SAEs that occur after the protocol-defined follow-up period has concluded and the event is deemed relevant to the use of study drug, the investigator should promptly document and report the event to Gilead PVE.

All AEs and SAEs will be recorded in the eCRF database within the timelines outlined in the eCRF completion guidelines.

### 7.3.3.1. Electronic Serious Adverse Event (eSAE) Reporting Process

• Site personnel record all SAE data on the applicable eCRFs and from there transmit the SAE information to Gilead PVE within 24 hours of the investigator's knowledge of the event. Detailed instructions can be found in the eCRF completion guidelines.

• If it is not possible to record and submit the SAE information electronically, because the eCRF database cannot be accessed or is not available (including at study-start), record the SAE on the paper SAE reporting form and submit within 24 hours to:

Gilead PVE
Email: PPD
or
Fax: PPD

- As soon as it is possible to do so, any SAE reported via paper must be transcribed on the applicable eCRFs according to instructions and within the timelines outlined in the eCRF completion guidelines.
- If an SAE has been reported via a paper form because the eCRF database has been locked, no further action is necessary.
- For fatal or life-threatening events, copies of hospital case reports, autopsy reports, and other documents are also to be submitted by email or fax when requested and applicable.
   Transmission of such documents should occur without personal subject identification, maintaining the traceability of a document to the subject identifiers.
- Additional information may be requested to ensure the timely completion of accurate safety reports.
- Any medications necessary for treatment of the SAE must be recorded onto the concomitant medication section of the subject's eCRF and the SAE narrative section of the Safety Report Form eCRF.

## 7.4. Gilead Reporting Requirements

Depending on relevant local legislation or regulations, including the applicable US FDA Code of Federal Regulations, the European Union (EU) Clinical Trials Directive (2001/20/EC) and relevant updates, and other country-specific legislation or regulations, Gilead may be required to expedite to worldwide regulatory agencies reports of SAEs, serious adverse drug reactions (SADRs), or suspected unexpected serious adverse reactions (SUSARs). In accordance with the EU Clinical Trials Directive (2001/20/EC), Gilead or a specified designee will notify worldwide regulatory agencies and the relevant IEC in concerned Member States of applicable SUSARs as outlined in current regulations.

Assessment of expectedness for SAEs will be determined by Gilead using reference safety information specified in the investigator's brochure or relevant local label as applicable.

All investigators will receive a safety letter notifying them of relevant SUSAR reports associated with any study drug. The investigator should notify the IRB or IEC of SUSAR reports as soon as is practical, where this is required by local regulatory agencies, and in accordance with the local institutional policy.

# 7.5. Clinical Laboratory Abnormalities and Other Abnormal Assessments as Adverse Events or Serious Adverse Events

Laboratory abnormalities without clinical significance are not recorded as AEs or SAEs. However, laboratory abnormalities (eg, clinical chemistry, hematology, and urinalysis) that require medical or surgical intervention or lead to study drug interruption, modification, or discontinuation must be recorded as an AE, as well as an SAE, if applicable. In addition, laboratory or other abnormal assessments (eg, electrocardiogram, x-rays, vital signs) that are associated with signs and/or symptoms must be recorded as an AE or SAE if they meet the definition of an AE or SAE as described in Sections 7.1.1 and 7.1.2. If the laboratory abnormality is part of a syndrome, record the syndrome or diagnosis (eg, anemia), not the laboratory result (ie, decreased hemoglobin).

Laboratory abnormalities that do not require medical intervention or action are generally not considered AEs.

Severity should be recorded and graded according to the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 dated July 2017. For AEs associated with laboratory abnormalities, the event should be graded on the basis of the clinical severity in the context of the underlying conditions; this may or may not be in agreement with the grading of the laboratory abnormality.

## 7.6. Special Situations Reports

#### 7.6.1. Definitions of Special Situations

Special situation reports include all reports of medication error, abuse, misuse, overdose, occupational exposure, drug interactions, exposure via breastfeeding, unexpected benefit, transmission of infectious agents via the product, counterfeit of falsified medicine, and pregnancy regardless of an associated AE.

Medication error is any unintentional error in the prescribing, dispensing, preparation for administration or administration of an investigational product while the medication is in the control of a health care professional, patient, or consumer. Medication errors may be classified as a medication error without an AE, which includes situations of missed dose; medication error with an AE; intercepted medication error; or potential medication error.

Abuse is defined as persistent or sporadic intentional excessive use of an investigational product by a subject.

Misuse is defined as any intentional and inappropriate use of an investigational product that is not in accordance with the protocol instructions or the local prescribing information.

An overdose is defined as an accidental or intentional administration of a quantity of an investigational product given per administration or cumulatively which is above the maximum recommended dose as per protocol or in the product labeling (as it applies to the daily dose of the subject in question). In cases of a discrepancy in drug accountability, overdose will be established only when it is clear that the subject has taken the excess dose(s). Overdose cannot be established when the subject cannot account for the discrepancy except in cases in which the investigator has reason to suspect that the subject has taken the additional dose(s).

Occupational exposure is defined as exposure to an investigational product as a result of one's professional or non-professional occupation.

Drug interaction is defined as any drug/drug, drug/food, or drug/device interaction.

Unexpected benefit is defined as an unintended therapeutic effect where the results are judged to be desirable and beneficial.

Transmission of infectious agents is defined as any suspected transmission of an infected agent through a Gilead investigational product.

Counterfeit or falsified medicine: Any investigational product with a false representation of: a) its identity, b) its source, or c) its history.

## 7.6.2. Instructions for Reporting Special Situations

### 7.6.2.1. Instructions for Reporting Pregnancies

The investigator should report pregnancies in female study subjects that are identified after initiation of study drug and throughout the study, including the post study drug follow-up period, to the Gilead PVE using the pregnancy report form within 24 hours of becoming aware of the pregnancy.

Gilead PVE
Email: PPD
or
Fax: PPD

Refer to Section 7.3 and the eCRF completion guidelines for full instructions on the mechanism of pregnancy reporting.

The pregnancy itself is not considered an AE nor is an induced elective abortion to terminate a pregnancy without medical reasons.

Any premature termination of pregnancy (eg, a spontaneous abortion, an induced therapeutic abortion due to complications or other medical reasons) must be reported within 24 hours as an SAE. The underlying medical reason for this procedure should be recorded as the AE term.

A spontaneous abortion is always considered to be an SAE and will be reported as described in Sections 7.3.3. Furthermore, any SAE occurring as an adverse pregnancy outcome post study must be reported to Gilead PVE.

The subject should receive appropriate monitoring and care until the conclusion of the pregnancy. The outcome should be reported to Gilead PVE using the pregnancy outcome report form. If the end of the pregnancy occurs after the study has been completed, the outcome should be reported directly to Gilead PVE. Gilead PVE contact information is as follows:

email: PPD and fax: PPD

Pregnancies of female partners of male study subjects exposed to Gilead or other study drugs must also be reported and relevant information should be submitted to Gilead PVE using the pregnancy and pregnancy outcome forms within 24 hours. If the end of the pregnancy occurs after the study has been completed, the outcome should be reported directly to Gilead PVE, fax number PPD or email PPD

Refer to Appendix 3 for Pregnancy Precautions, Definition for Female of Childbearing Potential, and Contraceptive Requirements.

## 7.6.2.2. Reporting Other Special Situations

All other special situation reports must be reported on the special situations report form and forwarded to the Gilead PVE within 24 hours of the investigator becoming aware of the situation. These reports must consist of situations that involve study drug and/or Gilead concomitant medications, but do not apply to non-Gilead concomitant medications.

Gilead PVE
Email: PPD
or
Fax: PPD

Special situations involving non-Gilead concomitant medications do not need to be reported on the special situations report form; however, special situations that result in AEs due to a non-Gilead concomitant medication, must be reported as an AE.

Any inappropriate use of concomitant medications prohibited by this protocol should not be reported as "misuse," but may be more appropriately documented as a protocol deviation.

Refer to Section 7.3 and the eCRF completion guidelines for instructions on special situation reporting.

All clinical sequelae in relation to these special situation reports will be reported as AEs or SAEs at the same time using the AE eCRF and/or the SAE report form. Details of the symptoms and signs, clinical management, and outcome will be reported, when available.

## 8. STATISTICAL CONSIDERATIONS

#### 8.1. Analysis Objectives and Endpoints

The purpose of this study is to provide RDV to participants with severe COVID-19.

### 8.1.1. Analysis Objectives

The analysis objectives of this study are as follows:

- To evaluate the efficacy of 2 RDV regimens with respect to clinical status assessed by a 7-point ordinal scale on Day 14
- To evaluate the safety and tolerability of RDV

## 8.1.2. Primary Endpoint

The primary endpoint of this study is:

• Clinical status assessed by a 7-point ordinal scale on Day 14

## 8.1.3. Secondary Endpoint

The secondary endpoint of this study is:

• The proportion of participants with treatment emergent AEs

## 8.1.4. Other Endpoints of Interest

Other endpoints of interest are:

- Time to  $SpO_2 > 94\%$  on room air
- Time to first negative SARS-CoV-2 PCR
- Duration of oxygen therapy (days)
- Duration of hospitalization (days)
- All cause mortality at Day 28
- Time to clinical improvement (days): Clinical improvement defined a ≥ 2-point improvement from Day 1 on a 7-point ordinal scale
- The proportion of participants in the Mechanically Ventilated Treatment Group and Extension Treatment Group with treatment-emergent AEs

## 8.2. Planned Analyses

## 8.2.1. Interim Analysis

Prior to the final analysis, the primary analysis of the primary endpoint will be conducted, additional interim analyses may be conducted, and the analyses may be submitted to regulatory agencies to seek guidance for the overall clinical development program or for other purposes.

### 8.2.1.1. DMC Analysis

The DMC will review safety and efficacy data on a regular basis.

#### 8.2.2. Primary Analysis

The primary analysis will be performed after all participants have completed 14 days in Part A of the study or prematurely terminated from Part A of the study prior to 14 days.

## 8.2.3. Final Analysis

The final analysis will be performed after all participants have completed the study or prematurely terminated from the study, outstanding data queries have been resolved or adjudicated as unresolvable, and the data have been cleaned and finalized.

## 8.3. Analysis Conventions

#### 8.3.1. Analysis Sets

#### 8.3.1.1. Efficacy

The primary analysis set for efficacy analysis is defined as the full analysis set (FAS), which will include all participants who (1) are randomized into Part A of the study and (2) have received at least 1 dose of RDV. Participants will be grouped according to the treatment to which they were randomized.

### 8.3.1.2. Safety

The primary analysis set for safety analyses is defined as the Safety Analysis Set, which will include all participants who (1) are randomized into the study and (2) have received at least 1 dose of RDV. Participants will be grouped according to the treatment to which they were randomized for Part A (5-day dosing group or 10-day dosing group) and according to the treatment to which they were assigned for Part B (Mechanically Ventilated Treatment Group or Extension Treatment Group).

## 8.3.1.3. Expanded RDV-Treated Analysis Set

The Expanded RDV-Treated Analysis Set will include participants who have received at least 1 dose of RDV in either the Mechanically Ventilated Treatment Group or Extension Treatment Group. This analysis set will be used for both the safety and efficacy evaluations for participants enrolled in Part B.

## 8.3.2. Data Handling Conventions



Laboratory data that are continuous in nature but are less than the lower limit of quantitation or above the upper limit of quantitation, will be imputed to the value of the lower or upper limit plus or minus 1 significant digit, respectively (eg, if the result of a continuous laboratory test is < 20, a value of 19 will be assigned).

Missing data can have an impact upon the interpretation of the trial data. In general, values for missing data will not be imputed. However, a missing pre-treatment laboratory result would be treated as normal (ie, no toxicity grade) for the laboratory abnormality summary.

All available data for participants that do not complete the study will be included in data listings

## 8.4. Demographic and Baseline Characteristics Analysis

Demographic and baseline measurements will be summarized using standard descriptive methods. Demographic summaries will include sex, race/ethnicity, and age. For categorical demographic and baseline characteristics, a Cochran Mantel Haenszel test will be used to compare treatment groups in Part A. For continuous demographic and baseline characteristics, a Wilcoxon rank sum test will be used to compare treatment groups in Part A.

### 8.5. Efficacy Analysis

## 8.5.1. Primary Analysis

The primary endpoint will be analyzed using a proportional odds model. The null hypothesis being tested is whether the odds of improvement on the ordinal scale is the same for the two treatment groups (ie, whether the common odds ratio is equal to 1). The odds ratio and 95% confidence interval will be provided.

The proportion of subjects in each category will be summarized by treatment group. The validity of the proportionality assumption will be evaluated.

If a participant is discharged prior to Day 14, the Day 14 ordinal scale category is considered to be not hospitalized. Every effort will be made to obtain clinical status data for all subjects prior to discharge. Subjects who have missing clinical status information on Day 14 will be excluded from the primary analysis.

### 8.5.2. Secondary Analyses

The secondary endpoint of proportion of participants with treatment emergent AEs will be compared between the 2 treatment groups in Part A using a Fisher's Exact test. The point estimate of the treatment difference and the associated 95% confidence intervals will be provided. Secondary or other endpoints of interest related to proportion of participants will be compared between treatment groups in Part A using a chi-square test or Fisher's Exact test. Endpoints that are measured as time to first event will be compared between treatment groups using the Log-Rank test and continuous endpoints will be compared between treatment groups using a Wilcoxon rank sum test or analysis of variance model.

For Part B, summaries of the 7-point scale ordinal scale and other efficacy endpoints of interest will be provided by group (Mechanically Ventilated Treatment Group or Extension Treatment Group).

## 8.6. Safety Analysis

All safety data collected on or after the date that study drug was first dispensed through the Day 28 follow-up visit will be summarized by treatment group (according to the study drug received). Data for the pretreatment period will be included in data listings.

Summaries will be provided by group: 5-day dosing group or 10-day dosing group for Part A and Mechanically Ventilated Treatment Group or Extension Treatment Group for Part B.

#### 8.6.1. Extent of Exposure

A subject's extent of exposure to study drug data will be generated from the study drug administration data. Exposure data will be summarized by group.

### **8.6.2.** Adverse Events

Clinical and laboratory AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). System Organ Class (SOC), High-Level Group Term (HLGT), High-Level Term (HLT), Preferred Term (PT), and Lower-Level Term (LLT) will be attached to the clinical database.

Events will be summarized on the basis of the date of onset for the event. A treatment-emergent AE will be defined as any AE that begins on or after the date of first dose of study drug up to the date of last dose of study drug plus 30 days, or up to Day 28, whichever is the later date.

Summaries (number and percentage of participants) of treatment-emergent AEs (by SOC, and PT) will be provided by group.

## 8.6.3. Laboratory Evaluations

Selected laboratory data will be summarized using only observed data. Data and change from baseline at all scheduled time points will be summarized.

Graded laboratory abnormalities will be defined using the grading scheme in DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Event, Version 2.1 dated July 2017.

Incidence of treatment-emergent laboratory abnormalities, defined as values that increase at least 1 toxicity grade from baseline at any time post baseline up to and including the date of last dose of study drug plus 30 days will be summarized by treatment group. If baseline data are missing, then any graded abnormality (ie, at least a Grade 1) will be considered treatment-emergent.

Laboratory abnormalities that occur before the first dose of study drug or after the subject has been discontinued from treatment for more than 30 days will be included in a data listing.



## 8.8. Adjustments for Multiplicity

No adjustments for multiple comparisons are planned.

### 8.9. Sample Size

The sample size computation is based on an assumed distribution of the 7-point ordinal scale on Day 14 for Part A Treatment Group 1. The odds ratio represents the odds of improvement in the ordinal scale for Treatment Group 2 relative to Treatment Group 1. The sample size needed to detect a given odds ratio for a 1:1 randomization using a 2-tailed test at level  $\alpha$  is given by:

12 
$$(z_{\alpha/2} + z_{\beta})^2 / \theta^2 (1 - \sum_{i=1}^{7} \rho_i^3)$$

Where  $\theta$  is the log odds ratio,  $\rho_i$  is the overall probability (combined over both treatment groups) of being in the ith category of the ordinal outcome, and  $z_{\alpha/2}$  and  $z_{\beta}$  are the 1-  $\alpha/2$  and  $\beta$  quantiles of the standard normal distribution {Whitehead 1993}.

A sample size of 400 participants (200 in each group) achieves > 85% power to detect an odds ratio of 1.75 using a two-sided significance level of 0.05. In this sample size calculation, it is assumed that the probability distribution of the ordinal scale at Day 14 for Group 1 is as follows:

- 1. Death, 2%
- 2. Hospitalized, on invasive mechanical ventilation or ECMO, 4%

- 3. Hospitalized, on non-invasive ventilation or high flow oxygen devices, 7%
- 4. Hospitalized, requiring low flow supplemental oxygen, 13%
- 5. Hospitalized, not requiring supplemental oxygen requiring ongoing medical care (COVID-19 related or otherwise), 16%
- 6. Hospitalized, not requiring supplemental oxygen no longer requires ongoing medical care (other than per protocol RDV administration), 20%
- 7. Not hospitalized, 38%

The sample size calculation was done using software PASS (Version 14.0).

## 8.10. Data Monitoring Committee

An external Independent Data Monitoring Committee (IDMC) includes independent experts that do not have direct involvement in the conduct of the study. The IDMC will review the progress of the study and perform interim reviews of safety data, and provide recommendation to Gilead whether the nature, frequency, and severity of adverse effects associated with study treatment warrant the early termination of the study in the best interests of the participants, whether the study should continue as planned, or the study should continue with modifications. The IDMC's specific activities will be defined by a mutually agreed charter, which will define the IDMC's membership, conduct and meeting schedule.

While the IDMC will be asked to advise Gilead regarding future conduct of the study, including possible early study termination, Gilead retains final decision-making authority on all aspects of the study.

## 9. **RESPONSIBILITIES**

### 9.1. Investigator Responsibilities

#### 9.1.1. Good Clinical Practice

The investigator will ensure that this study is conducted in accordance with ICH E6(R2) addendum to its guideline for GCP and applicable laws and regulations including the principles of the Declaration of Helsinki.

#### 9.1.2. Financial Disclosure

The investigator and subinvestigators will provide prompt and accurate documentation of their financial interest or arrangements with Gilead, or proprietary interests in the investigational drug during the course of a clinical study. This documentation must be provided prior to the investigator's (and any subinvestigator's) participation in the study. The investigator and subinvestigator agree to notify Gilead of any change in reportable interests during the study and for 1 year following completion of the study. Study completion is defined as the date when the last subject completes the protocol-defined activities.

# 9.1.3. Institutional Review Board/Independent Ethics Committee Review and Approval

The investigator (or Gilead as appropriate according to local regulations) will submit this protocol, informed consent form, and any accompanying material to be provided to the subject (such as advertisements, subject information sheets, or descriptions of the study used to obtain informed consent) to an IRB/IEC. The investigator will not begin any study subject activities until approval from the IRB/IEC has been documented and provided as a letter to the investigator.

Before implementation, the investigator will submit to and receive documented approval from the IRB/IEC any modifications made to the protocol or any accompanying material to be provided to the subject after initial IRB/IEC approval, with the exception of those necessary to reduce immediate risk to study subjects.

#### 9.1.4. Informed Consent (or Assent)

The investigator is responsible for obtaining written informed consent from the participant, or with a legal representative who can provide informed consent, or enrolled under ICH E6(R2) 4.8.15 emergency use provisions as deemed necessary by the investigator (participants  $\geq 18$  years of age), or obtaining or assent (age  $\geq 12$  to <18, where locally and nationally approved) from each individual participating in this study after adequate explanation of the aims, methods, objectives, and potential hazards of the study before undertaking any study-related procedures. The investigator must use the most current IRB- or IEC-approved consent form for documenting written informed consent. Each informed consent (or assent as applicable) will be appropriately

signed and dated by the subject or the subject's legally authorized representative and the person conducting the consent discussion, and also by an impartial witness if required by IRB or IEC or local requirements.

### 9.1.5. Confidentiality

The investigator must assure that subjects' anonymity will be strictly maintained and that their identities are protected from unauthorized parties. Only an identification code and any other unique identifier(s) as allowed by local law (such as year of birth) will be recorded on any form or biological sample submitted to Gilead, IRB or IEC. No biological samples will be provided to Gilead or any central laboratory during this study. NOTE: The investigator must keep a screening log with details for all subjects screened and enrolled in the study, in accordance with the site procedures and regulations. Subject data will be processed in accordance with all applicable regulations.

The investigator agrees that all information received from Gilead, including but not limited to the investigator's brochure, this protocol, CRF/eCRF, the study drug, and any other study information, remain the sole and exclusive property of Gilead during the conduct of the study and thereafter. This information is not to be disclosed to any third party (except employees or agents directly involved in the conduct of the study or as required by law) without prior written consent from Gilead. The investigator further agrees to take all reasonable precautions to prevent the disclosure by any employee or agent of the study site to any third party or otherwise into the public domain.

### 9.1.6. Study Files and Retention of Records

The investigator must maintain adequate and accurate records to enable the conduct of the study to be fully documented and the study data to be subsequently verified. These documents should be classified into at least the following 2 categories: (1) investigator's study file, and (2) subject clinical source documents.

The investigator's study file will contain the protocol/amendments, paper or electronic completed subject CRFs, IRB or IEC and governmental approval with correspondence, informed consent, drug records, staff curriculum vitae and authorization forms, and other appropriate documents and correspondence.

The required source data should include sequential notes containing at least the following information for each subject:

- Subject identification;
- Documentation that subject meets eligibility criteria, ie, medical history, physical examination, and confirmation of diagnosis (to support inclusion and exclusion criteria);
- Documentation of the reason(s) a consented subject is not enrolled;
- Participation in study (including study number);

- Study discussed and date of informed consent;
- Dates of all visits;
- Documentation that protocol-specific procedures were performed;
- Results of efficacy parameters, as required by the protocol;
- Start and end date (including dose regimen) of study drug, including dates of dispensing and return;
- Record of all AEs and other safety parameters (start and end date, and including causality and severity), and documentation that adequate medical care has been provided for any AE;
- Concomitant medication (including start and end date, dose if relevant; dose changes);
- Date of study completion and reason for early discontinuation, if it occurs.

All clinical study documents must be retained by the investigator until at least 2 years or according to local laws, whichever is longer, after the last approval of a marketing application in an ICH region (ie, US, Europe, or Japan) and until there are no pending or planned marketing applications in an ICH region; or, if no application is filed or if the application is not approved for such indication, until 2 years after the investigation is discontinued and regulatory authorities have been notified. Investigators may be required to retain documents longer if specified by regulatory requirements, by local regulations, or by an agreement with Gilead. The investigator must notify Gilead before destroying any clinical study records.

Should the investigator wish to assign the study records to another party or move them to another location, Gilead must be notified in advance.

If the investigator cannot provide for this archiving requirement at the study site for any or all of the documents, special arrangements must be made between the investigator and Gilead to store these records securely away from the site so that they can be returned sealed to the investigator in case of an inspection. When source documents are required for the continued care of the subject, appropriate copies should be made for storage away from the site.

### 9.1.7. Case Report Forms

For each subject consented, an eCRF casebook will be completed by an authorized study staff member whose training for this function is completed in the electronic data capture (EDC) system. The eCRF casebook will only capture the data required per the protocol schedule of events and procedures. The Inclusion/Exclusion Criteria and Enrollment eCRFs should be completed only after all data related to eligibility have been received. Data entry should be performed in accordance with the eCRF Completion Guidelines (eCCGs) provided by the Sponsor. Subsequent to data entry, a study monitor will perform source data verification (SDV) within the EDC system. System-generated or manual queries will be issued in the EDC system as data discrepancies are identified by the monitor or Gilead staff, who routinely review the data for completeness, correctness, and consistency. The site investigator or site coordinator or other

designee is responsible for responding to the queries in a timely manner, within the system, either by confirming the data as correct or updating the original entry, and providing the reason for the update (e.g. data entry error). Original entries as well as any changes to data fields will be stored in the audit trail of the system. At a minimum, prior to any interim time points or database lock (as instructed by Gilead), the investigator will use his/her log in credentials to confirm that the forms have been reviewed, and that the entries accurately reflect the information in the source documents. At the conclusion of the study, Gilead will provide the site investigator with a read-only archive copy of the data entered by that site. This archive must be stored in accordance with the records retention requirements outlined in Section 9.1.6.

## 9.1.8. Investigator Inspections

The investigator will make available all source documents and other records for this study to Gilead's appointed study monitors, to IRBs/IECs, or to regulatory authority or health authority inspectors.

## 9.1.9. Protocol Compliance

The investigator is responsible for ensuring the study is conducted in accordance with the procedures and evaluations described in this protocol.

## 9.2. Sponsor Responsibilities

#### 9.2.1. Protocol Modifications

Protocol modifications, except those intended to reduce immediate risk to study subjects, may be made only by Gilead. The investigator must submit all protocol modifications to the IRB/IEC in accordance with local requirements and receive documented IRB/IEC approval before modifications can be implemented.

## 9.2.2. Study Report and Publications

A clinical study report (CSR) will be prepared and provided to the regulatory agency(ies). Gilead will ensure that the report meets the standards set out in the ICH Guideline for Structure and Content of Clinical Study Reports (ICH E3). Note that an abbreviated report may be prepared in certain cases.

Investigators in this study may communicate, orally present, or publish in scientific journals or other scholarly media only after the following conditions have been met:

The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form or the study has been completed at all study sites for at least 2 years.

The investigator will submit to Gilead any proposed publication or presentation along with the respective scientific journal or presentation forum at least 30 days before submission of the publication or presentation.

No such communication, presentation, or publication will include Gilead's confidential information (see Section 9.1.5).

The investigator will comply with Gilead's request to delete references to its confidential information (other than the study results) in any paper or presentation and agrees to withhold publication or presentation for an additional 60 days in order to obtain patent protection if deemed necessary.

#### 9.3. Joint Investigator/Sponsor Responsibilities

## 9.3.1. Payment Reporting

Investigators and their study staff may be asked to provide services performed under this protocol, eg, attendance at Investigator Meetings. If required under the applicable statutory and regulatory requirements, Gilead will capture and disclose to Federal and State agencies any expenses paid or reimbursed for such services, including any clinical study payments, meal, travel expenses or reimbursements, consulting fees, and any other transfer of value.

## 9.3.2. Access to Information for Monitoring

The monitor is responsible for routine review of the CRF/eCRF at regular intervals throughout the study to verify adherence to the protocol and the completeness, consistency, and accuracy of the data being entered on them. The monitor should have access to any subject records needed to verify the entries in the CRF/eCRF. The investigator agrees to cooperate with the monitor to ensure that any problems detected through any type of monitoring (central, on site) are resolved.

#### 9.3.3. Access to Information for Auditing or Inspections

Representatives of regulatory authorities or of Gilead may conduct inspections or audits of the clinical study. If the investigator is notified of an inspection by a regulatory authority the investigator agrees to notify the Gilead medical monitor immediately. The investigator agrees to provide to representatives of a regulatory agency or Gilead access to records, facilities, and personnel for the effective conduct of any inspection or audit.

### 9.3.4. Study Discontinuation

Both Gilead and the investigator reserve the right to terminate the study at any time. Should this be necessary, both parties will arrange discontinuation procedures and notify the subjects, appropriate regulatory authorities, IRB/IECs. In terminating the study, Gilead and the investigator will assure that adequate consideration is given to the protection of the subjects' interests.

### 10. REFERENCES

- Cockcroft DW, Gault MH. Prediction of creatinine clearance from serum creatinine. Nephron 1976;16:31-41.
- De Wit E, Feldmann F, Cronin J, Jordan R, Okumura A, Thomas T, et al. Prophylactic and Therapeutic Remdesivir (GS-5734) Treatment in the Rhesus Macaque Model of MERS-CoV Infection. PNAS Latest Articles 2020.
- Sheahan TP, Sims AC, Graham RL, Menachery VD, Gralinski LE, Case JB, et al. Broad-Spectrum Antiviral GS-5734 Inhibits Both Epidemic and Zoonotic Coronaviruses. Science translational medicine 2017:1-20.
- Sheahan TP, Sims AC, Leist SR, Schafer A, Won J, Brown AJ, et al. Comparative Therapeutic Efficacy of Remdesivir and Combination Lopinavir, Ritonavir, and Interferon Beta Against MERS-CoV. Nature communications 2020;11:222.
- TAMIFLU®, Genentech Inc. TAMIFLU® (oseltamivir phosphate) capsules for oral use, TAMIFLU® (oseltamivir phosphate) for oral suspension. U.S. Prescribing Information. South San Francisco, CA. Revised August. 2019:
- Wang M, Cao R, Zhang L, Yang X, Liu J, Xu M, et al. Remdesivir and Chloroquine Effectively Inhibit the Recently Emerged Novel Coronavirus (2019-nCoV) In Vitro. Cell research 2020;30:269-71.
- Whitehead J. Sample size calculations for ordered categorical data. Stat Med 1993;12 (24):2257-71.
- World Health Organisation (WHO). Coronavirus Disease 2019 (COVID-19) Situation Report 34, 2020.

# 11. APPENDICES

Appendix 1. Investigator Signature Page Appendix 2. Study Procedures Table

Appendix 3. Pregnancy Precautions, Definition for Female of Childbearing Potential, and

Contraceptive Requirements

## Appendix 1. Investigator Signature Page

## GILEAD SCIENCES, INC. 333 LAKESIDE DRIVE FOSTER CITY, CA 94404

#### STUDY ACKNOWLEDGMENT

A Phase 3 Randomized Study to Evaluate the Safety and Antiviral Activity of Remdesivir (GS-5734<sup>TM</sup>) in Participants with Severe COVID-19 Protocol Amendment 3.0 12 April 2020 This protocol has been approved by Gilead Sciences, Inc. The following signature documents this approval. Signature 12 April 2020 Date INVESTIGATOR STATEMENT I have read the protocol, including all appendices, and I agree that it contains all necessary details for me and my staff to conduct this study as described. I will conduct this study as outlined herein and will make a reasonable effort to complete the study within the time designated. I will provide all study personnel under my supervision copies of the protocol and access to all information provided by Gilead Sciences, Inc. I will discuss this material with them to ensure that they are fully informed about the drugs and the study. Principal Investigator Name (Printed) Signature Date Site Number

## **Appendix 2.** Study Procedures Table

| | Screening | Baseline /<br>Day 1 <sup>b</sup> | Day 2 | Day 3 | Day 4 | Day 5 | Days 6<br>and 7 | Day 8 | Day 9 | Day 10 | Days 11,<br>12 and 13 | Day 14 | Day 28°<br>Follow-up<br>(±5 days) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Written Informed Consent | X | | | | | | | | | | | | |
| Medical History | X | | | | | | | | | | | | |
| Physical Examination | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Height | X | | | | | | | | | | | | |
| Vital Signs <sup>a</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Study Laboratory Testing | X | X | | X | | X | | X | | X | | X | |
| Respiratory Status | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Ordinal Scale | | X | X | X | X | X | X | X | X | X | X | X | X |
| Pregnancy Test | X | | | | | | | | | | | | |
| CCI | | | | | | | | | | | | | |
| RDV Dosing for Group 1 | | X | X | X | X | X | | | | | | | |
| RDV Dosing for Group 2 | | X | X | X | X | X | X | X | X | X | | | |
| Adverse Events | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Concomitant Medications | X | X | X | X | X | X | X | X | X | X | X | X | X |

a Includes heart rate, respiratory rate, temperature, blood pressure, SpO<sub>2</sub>, and body weight. Body weight collected on screening and Day 1 and otherwise if available.

b Assessments need not be repeated if performed within 24 hours of screening procedures; data collection other than adverse events should stop at Day 14 or discharge whichever is earlier.

Day 28 evaluations completed if the visit is conducted in person. Only AEs, ordinal scale, and concomitant medication review completed if visit conducted by phone.

# Appendix 3. Pregnancy Precautions, Definition for Female of Childbearing Potential, and Contraceptive Requirements

### 1) Definitions

## a. Definition of Childbearing Potential

For the purposes of this study, a female born subject is considered of childbearing potential following the initiation of puberty (Tanner stage 2) until becoming post-menopausal, unless permanently sterile or with medically documented ovarian failure. No documentation of Tanner stage will be required for people unless deemed prepubescent.

Women are considered to be in a postmenopausal state when they are  $\geq 54$  years of age with cessation of previously occurring menses for  $\geq 12$  months without an alternative cause. In addition, women of any age with amenorrhea of  $\geq 12$  months may also be considered postmenopausal if their follicle stimulating hormone (FSH) level is in the postmenopausal range and they are not using hormonal contraception or hormonal replacement therapy.

Permanent sterilization includes hysterectomy, bilateral oophorectomy, or bilateral salpingectomy in a female subject of any age. Tubal ligation is not considered a method of permanent sterilization for the purposes of this study.

## b. Definition of Male Fertility

For the purposes of this study, a male born subject is considered of fertile after the initiation of puberty unless permanently sterile by bilateral orchidectomy or medical documentation.

### 2) Contraception Requirements for Female Subjects

### a. Study Drug Effects on Pregnancy and Hormonal Contraception

Data from nonclinical studies of RDV have demonstrated no adverse effect on fertility or embryo-fetal development. Remdesivir has not yet been studied in pregnant women. Before enrolling into studies with RDV, women of childbearing potential must have pregnancy testing performed at screening.

Available data indicate that RDV potentially causes an interaction with hormonal contraception that is considered of limited significance. Hormonal methods must be used with a barrier method.

Please refer to the latest version of the IB for additional information.

## b. Contraception Requirements for Female Subjects of Childbearing Potential

The inclusion of female subjects of childbearing potential requires using at least an acceptable effective contraceptive measure. They must have a negative pregnancy test at screening. In the event of a delayed menstrual period (over 1 month between menstruations), a pregnancy test must be performed to rule out pregnancy. This is applicable also for women of childbearing potential with infrequent or irregular periods. They must also agree to 1 of the following from Screening until the last dose of the study drug:

• Complete abstinence from intercourse of reproductive potential. Abstinence is an acceptable method of contraception only when it is in line with the subject's preferred and usual lifestyle.

Or

• Consistent and correct use of 1 of the following methods of birth control listed below.

Non-hormonal intrauterine device (IUD)

Hormonal IUD (must be used with a barrier method)

Tubal sterilization

Vasectomy in the male partner (provided that the partner is the sole sexual partner and had confirmation of surgical success 3 months after procedure)

Barrier methods

- Female barriers: Diaphragm with spermicide or Cervical cap with spermicide
- Male barriers: Male condom (with or without spermicide)

Hormonal methods are restricted to drugs associated with the inhibition of ovulation. Each method must be used with a barrier method, preferably male condom. Hormonally-based contraceptives permitted for use in this protocol are as follows:

- Oral contraceptives (either combined or progesterone only)
- Injectable progesterone
- Subdermal contraceptive implant
- Transdermal contraceptive patch
- Contraceptive vaginal ring

Contraceptive methods must be locally approved to be permitted.

Female subjects must also refrain from egg donation and in vitro fertilization during treatment and until the last study drug dose.

Inclusion of methods of contraception in this list of permitted methods does not imply that the method is approved in any country or region. Methods should only be used if locally approved.

## 3) Contraception Requirements for Male Subjects

During the study male subjects with female partners of childbearing potential should use condoms when engaging in intercourse of reproductive potential.

## 4) Unacceptable Birth Control Methods

Birth control methods that are unacceptable include periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods), withdrawal (coitus interruptus), spermicides only, and lactational amenorrhea method (LAM). A Female condom and a male condom should not be used together.

### 5) Procedures to be Followed in the Event of Pregnancy

Subjects will be instructed to notify the investigator if they become pregnant at any time during the study. Subjects who become pregnant or who suspect that they are pregnant during the study must report the information to the investigator and discontinue study drug immediately. Subjects whose partner has become pregnant or suspects she is pregnant during the study must report the information to the investigator. Instructions for reporting pregnancy, partner pregnancy, and pregnancy outcome are outlined in Section 7.6.2.1.